CLINICAL TRIAL: NCT01355822
Title: Impact of the NO-donor Pentaerythrithyltetrantrate on Perinatal Outcome in High-risk Pregnancies: a Prospective Randomized Pilot Study
Brief Title: Impact of the NO-donor Pentaerythrithyltetrantrate on Perinatal Outcome in High-risk Pregnancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Prof. Dr. Ekkehard Schleußner, University Hospital Jena, Deartmet og Obstetrics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PETN_ESTG
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: High Risk Pregnancy
Keywords: abortion; perinatal death; IUGR; preterm birth; placental abruption; preeclampsia
MeSH Terms: conditions — Perinatal Death; Premature Birth; Abruptio Placentae; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo control
- PETN (Experimental): Pentalong, Actavis Germay: 80 mg twice a day
  Interventions: Drug: PETN

INTERVENTIONS:
Drug: PETN — Pentaerythrithyltetranitrate: 80 mg orally twice a day
  Other Names: Pentalong®, , Actavis Germany, Langenfeld, Germany
  Arms: PETN
Drug: Placebo control — orally, twice daily
  Arms: Placebo

SUMMARY:
Pregnancies resulting in IUGR and also in preeclampsia are strongly associated with typical underlying placental pathology revealing small placentas and maldevelopment of the decidual blood vessels, suggesting under-perfusion from the maternal circulation. Since nitric oxide (NO) donors can improve decreased uteroplacental perfusion without any negative effects on fetal circulation, these may prevent negative pregnancy outcomes in patients at risk.

The aim of this study is to evaluate the effectiveness of the long-lasting NO donor pentarythrithyltetranitrate (PETN) to reduce the likelihood of adverse pregnancy outcomes (intrauterine growth retardation / IUGR, perinatal death, placental abruption, and preterm delivery) in women recognized to be at risk for this outcome by abnormal uterine flow in mid gestation.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women 190 to 236 weeks of gestation
* abnormal uterine Doppler as defined by bilateral notching, unilateral notching and increased impedance with mean resistance index (RI) > 0.65 or with mean RI > 0.7 without notching at time of enrollement
* informed consent

Exclusion Criteria:

* multiple gestation
* documented chromosomal or major fetal abnormalities
* rupture of membranes and/or clinical chorioamnionitis at time of enrolment
* maternal disease defined as contraindication for intake of PETN

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2002-04; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of perinatal death and/or IUGR defined as birth weight below the 10th percentile | 19 -40 weeks of gestation

SECONDARY OUTCOMES:
Development of IUGR and severe IUGR defined as birth weight below the 5th percentile | 19-40 weeks of gestation
Preterm birth before completed 37 weeks of gestation and very early preterm birth before completed 32 weeks of gestation | 19 - 32 weeks of gestation
Development of preeclampsia | 19 - 40 weeks of gestation
Any form of placental abruption | 19 - 40 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Jena, Department of Obstetrics, Jena, Thuringia, Germany